CLINICAL TRIAL: NCT00968916
Title: An Open-label, Dose Escalation, Safety and Pharmacokinetics Phase 1 Study With AVE8062 Administered as a 30-minute Intravenous Infusion Every 3 Weeks in Patients With Advanced Solid Tumors.
Brief Title: Dose Escalation, Safety and Pharmacokinetic Study of AVE8062 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED10967
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — AC 7700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Level 1:
  15.5 mg/m2 of AVE8062 will be administered once in every 3 weeks, with 30-minute intravenous infusion and continued until unacceptable toxicity or disease progression or patient refusal
  Level 2:
  25 mg/m2 of AVE8062 will be administered once in every 3 weeks, with 30-minute intravenous infusion and continued until unacceptable toxicity or disease progression or patient refusal
  Level 3:
  35 mg/m2 of AVE8062 will be administered once in every 3 weeks, with 30-minute intravenous infusion and continued until unacceptable toxicity or disease progression or patient refusal
  Level 4:
  50 mg/m2 of AVE8062 will be administered once in every 3 weeks, with 30-minute intravenous infusion and continued until unacceptable toxicity or disease progression or patient refusal
  Interventions: Drug: ombrabulin (AVE8062)

INTERVENTIONS:
Drug: ombrabulin (AVE8062) — Pharmaceutical form: injection solution
  Route of administration: intravenous infusion

SUMMARY:
Primary objective: To determine the maximum tolerated dose based on the incidence of dose limiting toxicity and the maximum administered dose of AVE8062 administered every 3 weeks in patients with advanced solid tumors.

Secondary objectives:

* To assess the overall safety profile of the drug.
* To characterize the pharmacokinetic profile of AVE8062 and its active metabolite RPR 258063.
* To evaluate anti-tumor activity of the drug.

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 4-week screening phase, 21-day study treatment cycles, an end of treatment visit and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor that has become refractory to conventional treatment or for which no standard therapy exists.
* Patients with signed and dated Institutional Review Board (IRB)-approved patient informed consent form (ICF) prior to enrollment in the study.

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status > or = 2.
* Life expectancy of less than 12 weeks.
* Concurrent treatment with any other anticancer therapy, including chemotherapy, immunotherapy, radiotherapy, targeted therapy, gene therapy, or patients planning to receive these treatments during the study.
* Absence of histologically or cytologically proven cancer.
* Male patients who do not agree with contraception. Absence of negative serum/urinary pregnancy test within the 7 days prior to the enrollment in the study for female patients with childbearing potential. Patients must be post-menopausal, surgically sterile, or using "effective contraception" (the definition of "effective contraception" will be based on the judgment of the investigator).
* Washout period of less than 28 days from prior antitumor therapy (chemotherapy, targeted agents, immunotherapy and radiotherapy) or any investigational treatment, except for nitrosoureas, mitomycin which may not be used up to 42 days prior to the first cycle. No washout period is required for hormonal therapy, however, it must be discontinued before the first cycle.
* Not recovered from all previous therapies (radiation, surgery, and medications). Adverse events related to previous therapies must be National Cancer Institute Common Terminology Criteria grade < or = 1 (or alopecia < or = grade 2) at screening or returned to the subject's baseline prior to their most recent previous therapy.
* Symptomatic brain metastases and carcinomatous leptomeningitis.
* Other serious illness or medical conditions:

  * Existence of significant neurologic or psychiatric disorders impairing the ability to obtain consent.
  * Active infection.
  * Other serious illness not controlled by adequate treatment.
* Inadequate organ function including:

  * Absolute neutrophils counts<1.5 x 10^9/L
  * Platelets counts<100 x 10^9/L
  * Hemoglobin<9.0 g/dL (without red blood cells transfusion during 28 days prior to the test)
  * Calculated creatinin clearance<60 ml/min
  * Total bilirubin > or = 1.5 mg/dL
  * Alanine aminotransferase/aspartate aminotransferase>1.5 times the upper normal limits of the institutional norms.
  * Alkaline phosphatase (AP)>2.5 times the upper normal limits of the institutional norms. An increase of AP up to grade 2 would be accepted only if this increase is related to the presence of bone metastases. Bone specific isoenzyme AP should be greater than the pathological limit defined by the manufacturer as a sign of bone metastases.
* Documented medical history of myocardial infarction, documented angina pectoris, arrhythmia especially severe conduction disorder such as second or third degree atrio-ventricular block, stroke, or history of arterial or venous thrombo-embolism within the past 180 days requiring anticoagulants.
* Patient with a left ventricular ejection fraction<50% by echocardiography.
* Patient with a baseline QTc interval of >0.45, or family history of Long QT Syndrome
* Patient with uncontrolled hypertension and patient with organ damage related to hypertension such as left ventricular hypertrophy or grade 2 ocular funduscopic changes or kidney impairment.
* Patient with growing vessel disease (eg age-related macular degeneration, diabetic retinopathy, rheumatoid arthritis), or ongoing wound healing process. Patient should be enrolled in the study at least 28 days after surgery.
* 12-lead Electrocardiogram: ST- and T-wave changes suggesting ischemia
* Hypertension defined as systolic blood pressure (BP)>140 mmHg or diastolic BP>90 mmHg on two repeated measurements at 30 minutes intervals.
* Patient with one or more episodes of ventricular tachycardia with 3 or more consecutive premature beats, with a frequency > or = 180 beats/min.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity at Cycle 1 | 21 days

SECONDARY OUTCOMES:
Global safety profile based on treatment emergent adverse events, serious adverse events, and laboratory abnormalities | all cycles
Pharmacokinetic parameters of AVE8062: Cmax, AUC, CL, Vss, and t1/2 | Day 1 and 2 of Cycle 1, and day 1 of subsequent cycles
Pharmacokinetic parameters of AVE8062's active metabolite RPR258063: Cmax, AUC, t1/2, and Metabolic ratio | Day 1 and 2 of Cycle 1, and day 1 of subsequent cycles
Objective tumor response as defined by the Response Evaluation Criteria in Solid Tumors in evaluable patients | from patient informed consent to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Sanofi-Aventis Investigational Site Number 392002, Osaka Sayama-Shi
  - Sanofi-Aventis Investigational Site Number 392001, Sunto-Gun

REFERENCES:
- [Derived] Murakami H, Kurata T, Onozawa Y, Watanabe J, Ono A, Takahashi T, Yamamoto N, Fujisaka Y, Kiyota H, Hayashi H, Tanaka K, Nakagawa K, Kuroda S. An open-label, dose-escalation, safety, and pharmacokinetics phase I study of ombrabulin, a vascular disrupting agent, administered as a 30-min intravenous infusion every 3 weeks in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Mar;73(3):623-30. doi: 10.1007/s00280-014-2388-x. Epub 2014 Jan 30. PMID 24477603